CLINICAL TRIAL: NCT05849402
Title: Accelerated Intermittent Theta-Burst Stimulation (aiTBS) in Treatment-Resistant Depression of Bipolar II Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Bora Kim, Principal Investigator: Nolan Williams, MD, Stanford University / Protocol Director: Bora Kim, MD, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49486-RCT
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Bipolar II Disorder, Most Recent Episode Major Depressive; Current Depressive Episode; Treatment Resistant Depression
Keywords: Bipolar II Disorder; Treatment Resistant Depression; Transcranial Magnetic Stimulation (TMS); Theta Burst
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active aiTBS (Active Comparator): Participants will be randomized to active or sham aiTBS condition, and receive 10 aiTBS to left DLPFC (LDLPFC) sessions a day for 5 days of course.
  Interventions: Device: Active Comparator: Active aiTBS
- Sham aiTBS (Sham Comparator): Participants will be randomized to active or sham aiTBS condition, and receive 10 aiTBS to left DLPFC (LDLPFC) sessions a day for 5 days of course.
  Interventions: Device: Sham Comparator: Sham aiTBS

INTERVENTIONS:
Device: Active Comparator: Active aiTBS — Participants will be randomized to active or sham aiTBS condition, and receive 10 aiTBS to left DLPFC (LDLPFC) sessions a day for 5 days of course.
  Arms: Active aiTBS
Device: Sham Comparator: Sham aiTBS — Participants will be randomized to active or sham aiTBS condition, and receive 10 aiTBS to left DLPFC (LDLPFC) sessions a day for 5 days of course.
  Arms: Sham aiTBS

SUMMARY:
The purpose of this study is to investigate the effectiveness of accelerated intermittent theta-burst transcranial magnetic stimulation (aiTBS) in inducing anti-depressant responses in individuals with treatment-resistant depression of bipolar II disorder. This is a double-blind, randomized, sham-controlled trial that targets a single location on the left dorsolateral prefrontal cortex (LDLPFC) using the MagPro rTMS system.

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy of aiTBS applied to the left dorsolateral prefrontal cortex (L-DLPFC) in reducing depressive symptoms in individuals with bipolar II disorder, and to determine the neural functional connectivity changes that underlie treatment response. A total of 60 individuals with bipolar II disorder who are currently experiencing a depressive episode will be recruited for the study.

The accelerated iTBS (aiTBS) treatment will consist of 10 sessions, administered daily over a period of 5 consecutive days. Before and after the stimulation, magnetic resonance imaging (MRI) scans, electroencephalograms (EEG), and heart rate variability (HRV) will be collected. The severity of depressive symptoms will be evaluated using both clinician-rated and self-report assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years old to 80 years old with a primary diagnosis of bipolar affective disorder II in a current major depressive episode, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Fourth Edition, Text Revision (DSM-V).
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
3. Meet the criteria by Maudsley Staging Method score >=7
4. Not in a current state of hypomania (as assessed by the Young Mania Rating Scale) or psychosis
5. In good general health, as ascertained by medical history.
6. Must have a stable psychiatrist during study enrollment, who confirms diagnosis of bipolar II disorder.
7. Must be on a mood stabilizer regimen for 6 weeks prior to study enrollment and agree to continue this regimen during study period
8. Meet the threshold on the MADRS, with a total score of >/=20 at screening/baseline.
9. TMS Naive

11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.

12. Agreement to adhere to Lifestyle Considerations throughout study duration.

Lifestyle considerations:

1. Abstain from becoming pregnant from the screening visit (Visit 1) until after the final study visit (Visit 9).
2. Continue usual intake patterns of caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) without significant change for the duration of the study.
3. Abstain from alcohol for at least 24 hours before the start of each MRI and TMS session.

Participants who use tobacco products will be informed that use will be allowed only in between intervention sessions.

Exclusion Criteria:

1. Primary diagnosis other than bipolar II disorder
2. Any structural lesion e.g. structural neurological condition, more subcortical lesions than would be expected for age, stroke effecting stimulated area or connected areas or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results.
3. Metal implant in brain (e.g. deep brain stimulation), cardiac pacemaker, or cochlear implants
4. History of epilepsy or seizures
5. Shrapnel or any ferromagnetic item in the head
6. Pregnancy
7. Autism Spectrum disorder
8. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation
9. Active substance abuse (<1 week) or intoxication verified by toxicology screen--of cocaine, amphetamines, benzodiazepines
10. Cognitive impairment (including dementia)
11. Current severe insomnia (must sleep a minimum of 5 hours the night before stimulation)
12. Current hypomania or psychosis
13. Showing symptoms of withdrawal from alcohol or benzodiazepines
14. A diagnosis of intellectual disability
15. Parkinsonism or other movement disorder determined by Principal Investigator to interfere with treatment
16. Any other indication the Principal Investigator feels would comprise data.
17. Current active suicidal ideation or suicide attempt or suicidal behaviors in the last 6 months
18. Any history of psycho surgery for depression
19. Any history of ECT (greater than 8 sessions) without meeting responder criteria
20. Recent (within 4 weeks of any clinical effect) or concurrent use of rapid acting antidepressant agent (i.e., ketamine or a course of ECT)

22. Any history of myocardial infarction, CABG, CHF, or other cardiac history

23. The presence or diagnosis of prominent anxiety disorder, personality disorder or dysthymia

24. History of intractable migraine

25. Hypomania in the past 6 months.

26. Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO)

27. Unstable symptoms between screening and baseline as defined by a 30% change in MADRS-C score.

28. Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Montgomery Asberg Depression Rating Scale (MADRS) | Baseline and immediately post-treatment, 1-month
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  The MADRS uses a 0 to 6 severity scale, scored following the interview. Scoring/Interpretation: Higher scores indicate increasing depressive symptoms. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.

SECONDARY OUTCOMES:
Change from baseline Young Mania Rating Scale (YMRS) | Baseline and immediate post-treatment, 1-month
  The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition.
  There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients.
  Typical YMRS baseline scores can vary a lot. They depend on the patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2).
Change in resting-state functional connectivity | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  Resting-state fMRI scans will be conducted before and after the course of aiTBS to examine changes in resting-state functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University; Bora Kim, MD, Study Director — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
www.clinicaltrials.gov

REFERENCES:
- [Background] Abraham WC, Bear MF. Metaplasticity: the plasticity of synaptic plasticity. Trends Neurosci. 1996 Apr;19(4):126-30. doi: 10.1016/s0166-2236(96)80018-x. PMID 8658594
- [Background] Baldessarini RJ, Tondo L, Davis P, Pompili M, Goodwin FK, Hennen J. Decreased risk of suicides and attempts during long-term lithium treatment: a meta-analytic review. Bipolar Disord. 2006 Oct;8(5 Pt 2):625-39. doi: 10.1111/j.1399-5618.2006.00344.x. PMID 17042835
- [Background] Beam W, Borckardt JJ, Reeves ST, George MS. An efficient and accurate new method for locating the F3 position for prefrontal TMS applications. Brain Stimul. 2009 Jan;2(1):50-4. doi: 10.1016/j.brs.2008.09.006. PMID 20539835
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Carpenter LL, Janicak PG, Aaronson ST, Boyadjis T, Brock DG, Cook IA, Dunner DL, Lanocha K, Solvason HB, Demitrack MA. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of acute treatment outcomes in clinical practice. Depress Anxiety. 2012 Jul;29(7):587-96. doi: 10.1002/da.21969. Epub 2012 Jun 11. PMID 22689344
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Geddes JR, Miklowitz DJ. Treatment of bipolar disorder. Lancet. 2013 May 11;381(9878):1672-82. doi: 10.1016/S0140-6736(13)60857-0. PMID 23663953
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Gibbons RD, Hedeker D, DuToit S. Advances in analysis of longitudinal data. Annu Rev Clin Psychol. 2010;6:79-107. doi: 10.1146/annurev.clinpsy.032408.153550. PMID 20192796
- [Background] Grisaru N, Chudakov B, Yaroslavsky Y, Belmaker RH. Transcranial magnetic stimulation in mania: a controlled study. Am J Psychiatry. 1998 Nov;155(11):1608-10. doi: 10.1176/ajp.155.11.1608. PMID 9812128
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Judd LL, Akiskal HS, Schettler PJ, Coryell W, Maser J, Rice JA, Solomon DA, Keller MB. The comparative clinical phenotype and long term longitudinal episode course of bipolar I and II: a clinical spectrum or distinct disorders? J Affect Disord. 2003 Jan;73(1-2):19-32. doi: 10.1016/s0165-0327(02)00324-5. PMID 12507734
- [Background] Leverich GS, Altshuler LL, Frye MA, Suppes T, McElroy SL, Keck PE Jr, Kupka RW, Denicoff KD, Nolen WA, Grunze H, Martinez MI, Post RM. Risk of switch in mood polarity to hypomania or mania in patients with bipolar depression during acute and continuation trials of venlafaxine, sertraline, and bupropion as adjuncts to mood stabilizers. Am J Psychiatry. 2006 Feb;163(2):232-9. doi: 10.1176/appi.ajp.163.2.232. PMID 16449476
- [Background] Li BJ, Friston K, Mody M, Wang HN, Lu HB, Hu DW. A brain network model for depression: From symptom understanding to disease intervention. CNS Neurosci Ther. 2018 Nov;24(11):1004-1019. doi: 10.1111/cns.12998. Epub 2018 Jun 21. PMID 29931740
- [Background] Merikangas KR, Jin R, He JP, Kessler RC, Lee S, Sampson NA, Viana MC, Andrade LH, Hu C, Karam EG, Ladea M, Medina-Mora ME, Ono Y, Posada-Villa J, Sagar R, Wells JE, Zarkov Z. Prevalence and correlates of bipolar spectrum disorder in the world mental health survey initiative. Arch Gen Psychiatry. 2011 Mar;68(3):241-51. doi: 10.1001/archgenpsychiatry.2011.12. PMID 21383262
- [Background] Miller S, Dell'Osso B, Ketter TA. The prevalence and burden of bipolar depression. J Affect Disord. 2014 Dec;169 Suppl 1:S3-11. doi: 10.1016/S0165-0327(14)70003-5. PMID 25533912
- [Background] Nyffeler T, Cazzoli D, Hess CW, Muri RM. One session of repeated parietal theta burst stimulation trains induces long-lasting improvement of visual neglect. Stroke. 2009 Aug;40(8):2791-6. doi: 10.1161/STROKEAHA.109.552323. Epub 2009 Jun 11. PMID 19520986
- [Background] Pascual-Leone A, Valls-Sole J, Brasil-Neto JP, Cammarota A, Grafman J, Hallett M. Akinesia in Parkinson's disease. II. Effects of subthreshold repetitive transcranial motor cortex stimulation. Neurology. 1994 May;44(5):892-8. doi: 10.1212/wnl.44.5.892. PMID 8190293
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Praharaj SK, Ram D, Arora M. Efficacy of high frequency (rapid) suprathreshold repetitive transcranial magnetic stimulation of right prefrontal cortex in bipolar mania: a randomized sham controlled study. J Affect Disord. 2009 Oct;117(3):146-50. doi: 10.1016/j.jad.2008.12.020. Epub 2009 Jan 28. PMID 19178948
- [Background] Rachid F, Moeglin C, Sentissi O. Repetitive Transcranial Magnetic Stimulation (5 and 10 Hz) With Modified Parameters in the Treatment of Resistant Unipolar and Bipolar Depression in a Private Practice Setting. J Psychiatr Pract. 2017 Mar;23(2):92-100. doi: 10.1097/PRA.0000000000000213. PMID 28291034
- [Background] Rostami R, Kazemi R, Nitsche MA, Gholipour F, Salehinejad MA. Clinical and demographic predictors of response to rTMS treatment in unipolar and bipolar depressive disorders. Clin Neurophysiol. 2017 Oct;128(10):1961-1970. doi: 10.1016/j.clinph.2017.07.395. Epub 2017 Jul 24. PMID 28829979
- [Background] Saba G, Rocamora JF, Kalalou K, Benadhira R, Plaze M, Lipski H, Januel D. Repetitive transcranial magnetic stimulation as an add-on therapy in the treatment of mania: a case series of eight patients. Psychiatry Res. 2004 Sep 30;128(2):199-202. doi: 10.1016/j.psychres.2004.05.019. PMID 15488963
- [Background] Thase ME. Bipolar depression: issues in diagnosis and treatment. Harv Rev Psychiatry. 2005 Sep-Oct;13(5):257-71. doi: 10.1080/10673220500326425. PMID 16251165
- [Background] Tondo L, Isacsson G, Baldessarini R. Suicidal behaviour in bipolar disorder: risk and prevention. CNS Drugs. 2003;17(7):491-511. doi: 10.2165/00023210-200317070-00003. PMID 12751919
- [Background] Tondo L, Vazquez G, Baldessarini RJ. Mania associated with antidepressant treatment: comprehensive meta-analytic review. Acta Psychiatr Scand. 2010 Jun;121(6):404-14. doi: 10.1111/j.1600-0447.2009.01514.x. Epub 2009 Dec 2. PMID 19958306